CLINICAL TRIAL: NCT05337072
Title: The FLORA-project: in Search for the Microbial Cause of Chronic Endometritis and the Most Appropriate Treatment to Obtain a Successful Pregnancy IVF/ICSI
Acronym: FLORA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Thomas Demuyser, Microbiologist, Universitair Ziekenhuis Brussel
Other Study IDs: FLORA-project
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Endometritis; Chronic; Subfertility
Keywords: Microbiome
MeSH Terms: conditions — Endometritis; Bronchiolitis Obliterans Syndrome; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swab Endometrial biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Microbiome study — Investigation of the vaginal and endometrial microbiome

SUMMARY:
Chronic endometritis is an inflammatory condition of the endometrium. This inflammation can negatively affect fertility and pregnancy. The pathology is frequently (+-10%) observed in women with fertility problems. Today, diagnosis of chronic endometritis is not evident, since no well-validated classification scales are available. In the UZ Brussel the pathology department applies its own in-house scoring system, based on the presence and position of plasma cells within the histological images.

Despite limited research so far, it recently became clear that the endometrium is colonized by micro-organisms (the microbiome). However, it is still unclear what role these microorganisms play in chronic endometritis and fertility problems. Chronic endometritis is often diagnosed in the context of fertility problems, and the patient is treated 'blindly' with broad-spectrum antibiotics such as doxycycline. Broad-spectrum antibiotics unnecessarily eradicate many microorganisms in our body, including the ones that positively influence implantation. The exact cause of chronic endometritis is unknown, so treatment remains empirical. The research and knowledge in the endometrial microbiome is constantly expanding, mainly due to the rise of research into the links between pathologies and human microbiota. It is becoming increasingly clear that the composition of the microbiome can play a vital role in health and disease. Regarding the influence of the endometrial microbiome on different pathologies, such as chronic endometritis and implantation failure or miscarriage, there is still no consensus. Despite multiple studies on the endometrial microbiome, we are not yet able to define a normal or healthy endometrial microbiome.

In this project, we want to gain insight into the microorganisms that are present in the female reproductive tract based on various techniques. The analyses will performed on an endometrial biopsy and a vaginal swab. The biopsy is routinely taken at Brussels IVF for the detection of plasma cells in the anatomopathology lab for the diagnosis of chronic endometritis. In the microbiology lab we will investigate which microorganisms are present in the female reproductive tract with and without the histological diagnosis of chronic endometritis. This will be done based on the state-of-the-art analytical techniques metagenomics (sequencing) and culturomics (culture).

DETAILED DESCRIPTION:
Chronic endometritis is an inflammatory condition of the endometrium. This inflammation can negatively affect fertility and pregnancy. The pathology is frequently (+-10%) observed in women with fertility problems. Today, diagnosis of chronic endometritis is not evident, since no well-validated classification scales are available. In the UZ Brussel the pathology department applies its own in-house scoring system, based on the presence and position of plasma cells within the histological images.

Despite limited research so far, it recently became clear that the endometrium is colonized by micro-organisms (the microbiome). However, it is still unclear what role these microorganisms play in chronic endometritis and fertility problems. Chronic endometritis is often diagnosed in the context of fertility problems, and the patient is treated 'blindly' with broad-spectrum antibiotics such as doxycyclin. Broad-spectrum antibiotics unnecessarily eradicate many microorganisms in our body, including the ones that positively influence implantation. The exact cause of chronic endometritis is unknown, so treatment remains empirical. The research and knowledge in the endometrial microbiome is constantly expanding, mainly due to the rise of research into the links between pathologies and human microbiota. It is becoming increasingly clear that the composition of the microbiome can play a vital role in health and disease. Regarding the influence of the endometrial microbiome on different pathologies, such as chronic endometritis and implantation failure or miscarriage, there is still no consensus. Despite multiple studies on the endometrial microbiome, we are not yet able to define a normal or healthy endometrial microbiome.

In this project, we want to gain insight into the microorganisms that are present in the female reproductive tract based on various techniques. The analyses will performed on an endometrial biopsy and a vaginal swab. The biopsy is routinely taken at Brussels IVF for the detection of plasma cells in the anatomopathology lab for the diagnosis of chronic endometritis. In the microbiology lab we will investigate which microorganisms are present in the female reproductive tract with and without the histological diagnosis of chronic endometritis. This will be done based on the state-of-the-art analytical techniques metagenomics (sequencing) and culturomics (culture)*. With metagenomics we detect genetic material of the micro-organisms directly in the samples, with culturomics we grow as many species as possible from the samples using a complex culture schedule, after which we identify these microorganisms using mass spectrometry. Culturomics is a new technique that has already been applied with great success abroad on various sample types resulting in the discovery of many new bacterial species. This technique has never been applied to vaginal swabs/endometrial biopsies, making it a very innovative project. The techniques culturomics and metagenomics are complementary to each other in obtaining a very complete picture of the microbiome.

It will be evaluated whether the microbiome of endometrial biopsies and vaginal swabs can offer help in the choice of an appropriate antibiotic when chronic endometritis is diagnosed in a patient. We will evaluate the microbiome at baseline and before and after treatment with (broad-spectrum) antibiotics, currently the first-choice being doxycyclin. We will examine what effect the antibiotic treatment has on the composition of the microbiome, to what extent the balance between "good and bad" bacteria has been restored and whether the histological signs (plasma cells) of chronic endometritis disappear.

The microbiological results will be compared to the classification score based on the presence of plasma cells. In this way, this unique classification score, which was developed in the anatomopathology laboratory of UZ Brussel, can be validated. Based on this classification score, a robust diagnosis is possible for a disease for which no substantiated diagnosis is available to date.

ELIGIBILITY:
Inclusion Criteria:

* Women planned for IVF/ICSI treatment at Brussels IVF (UZ Brussel)
* Women who undergo a diagnostic hysteroscopy in preparation of their treatment

Exclusion criteria:

* If an interventional instead of a diagnostic hysteroscopy in planned
* In the occurence If a previous history of chronic endometritis and the use of antibiotics in the last 3 months.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will include women planned for IVF/ICSI treatment at Brussels IVF (UZ Brussel) who undergo a diagnostic hysteroscopy in preparation of their treatment.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome analysis through sequencing and culture | 2 years
  The vaginal and endometrial microbiome will be evaluated through metagenomics sequencing and high-troughput culturomics.
  Metagenomics:
  An amplicon sequencing technique will be applied. Deep-sequencing metagenomic analysis will be performed. Microbiome bioinformatics and statistical data analyses will be performed through Quantitative Insights Into Microbial Ecology - QIIME2®. Community composition, biodiversity, and statistically different abundant taxa will be identified using appropriate statistical models, and visualisation methods.
  Culturomics:
  Two different pre-incubation conditions will be applied. We enrich both an aerobic and an anaerobic bloodculture bottle with sterile rumen fluid, sterile defibrinated sheep blood and a homemade supplement mix. Eight different agar plates will be used. After five days of incubation, all different bacterial and fungal colonies will be isolated for MALDI-TOF MS or 16S rRNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://researchportal.vub.be/nl/prizes/uz-brussel-foundation-flora-project-75-000